CLINICAL TRIAL: NCT01893489
Title: Phase I Study to Evaluated the Safety of Noninvasive Molecular Imaging for the Detection of Inflammation in Carotid Atherosclerotic Lesions by Using Ga-68-NOTA-MSA in Healthy Volunteers and Patients With Coronary Artery Disease
Brief Title: Visualization of Carotid Atherosclerosis by 68Ga-MSA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University (Other)
Collaborators: SHIN JIN MEDICS (Unknown)
Responsible Party: Principal Investigator, Hong Seog Seo, Professor of Medicine, Korea University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Ga_MSA_CAD_carotid
Record Dates: First submitted 2013-06-27; First posted 2013-07-09 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Atherosclerosis; Carotid Atherosclerosis; Noninvasive Imaging of Atherosclerosis
Keywords: positron emission tomography; macrophage; neomannosyl human serum albumin
MeSH Terms: conditions — Atherosclerosis; Carotid Artery Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atherosclerosis (Active Comparator): coronary artery disease patients with carotid plaques confirmed by a ultrasound study
  Interventions: Other: 68Gallium-MSA
- control (Sham Comparator): no coronary artery disease patients without carotid plaques confirmed by a ultrasound study
  Interventions: Other: 68Gallium-MSA

INTERVENTIONS:
Other: 68Gallium-MSA — 68Gallium-MSA 2.0 mci for Positron Emission Tomogram(PET) imaging

SUMMARY:
Until now, no specific atherosclerosis-targeting agent labeled with positron emitter is not yet available. Investigators developed neomannosyl human serum albumin(MSA) for the terminal mannose residues of MSA binding with the mannose receptors of macrophages in atherosclerosis, and investigators investigate whether 68Ga-MSA can be a novel agent for non-invasive molecular imaging of carotid atherosclerotic lesion in PET.

ELIGIBILITY:
Inclusion Criteria:

* •coronary artery disease patients with carotid plaques

  * control without carotid plaque

Exclusion Criteria:

* •pregnancy, allergy to albumin, any acute or chronic inflammatory disease, hematologic disease, liver disease, renal disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
side reactions at MSA injection site of the skin | with 2 hours after MSA injection
  development of unexpected skin rashes or other skin lesions at MSA injection site of the skin with 2 hours after MSA injection
unstable changes of vital signs and development of abnormal biochemical parameters | 24 hours after MSA injection
  This includes unstable changes of vital signs including blood pressure, body temperature and heart rate, and abnormal changes of biochemical parameters such as hematologic, hepatic and renal functions.

SECONDARY OUTCOMES:
standard uptake unit(SUV) at carotid arteries | baseline
SUV at aorta and iliac arteries | baseline

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Department of Nuclear Medicine, Institute of Radiation Medicine,, Seoul
  - Korea University Guro Hospital, Seoul